CLINICAL TRIAL: NCT00380588
Title: A Randomized Study of Gemcitabine/Cisplatin Versus Single-Agent Gemcitabine in Patients With Biliary Tract Cancer
Brief Title: Randomized Phase 2 Study With Gemcitabine Alone and Combination Therapy for Patients With Advanced Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10298; B9E-JE-BT22
Record Dates: First submitted 2006-09-22; First posted 2006-09-26 (Estimated); Results first posted 2009-11-19 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemcitabine + Cisplatin (Experimental): Gemcitabine: 1000 milligrams per square meter (mg/m2), intravenous (IV), day 1 and day 8 every 21 days x 16 maximum cycles or disease progression or unacceptable toxicity or patient withdrawal.
  Cisplatin: 25 milligrams per square meter (mg/m2), intravenous (IV), day 1 and day 8 every 21 days x 16 maximum cycles or disease progression or unacceptable toxicity or patient withdrawal.
  Interventions: Drug: gemcitabine; Drug: cisplatin
- Gemcitabine (Experimental): Gemcitabine: 1000 milligrams per square meter (mg/m2), intravenous (IV), day 1,8 and 15 every 28 days x 12 maximum cycles or disease progression or unacceptable toxicity or patient withdrawal.
  Interventions: Drug: gemcitabine

INTERVENTIONS:
Drug: gemcitabine — 1000 milligrams per square meter (mg/m2), intravenous (IV)
  Other Names: LY188011; Gemzar
Drug: cisplatin — 25 milligrams per square meter (mg/m2), intravenous (IV)
  Arms: Gemcitabine + Cisplatin

SUMMARY:
To investigate efficacy and safety of gemcitabine combined with cisplatin and of gemcitabine alone by comparison in patients with advanced biliary tract cancer

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of biliary tract cancer
* Measurable disease must be at least one lesion
* Chemotherapy-naïve
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Estimated life expectancy no less than 3 months

Exclusion Criteria:

* radiological or clinical evidence of pulmonary fibrosis or interstitial pneumonia

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2006-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- Japan (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine + Cisplatin | Gemcitabine
Started | 42 | 42
Received at Least One Dose of Study Drug | 41 | 42
Completed | 3 (Treatment period reached 48 week maximum.) | 2 (Treatment period reached 48 week maximum.)
Not Completed | 39 | 40
Not completed — Unequivocal Disease Progression | 25 | 34
Not completed — Next Cycle Not Started | 4 | 0
Not completed — Adverse Event | 7 | 3
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine + Cisplatin | Gemcitabine | Total
Number analyzed (Participants) | 41 | 42 | 83
Age Continuous [Mean (Standard Deviation); unit: years] | 63.7 (10.1) | 67.0 (6.9) | 65.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 44
  Male | 18 | 21 | 39
Region of Enrollment [Number; unit: participants]
  Japan | 41 | 42 | 83
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully Active | 34 | 28 | 62
    1 - Ambulatory, Restricted Strenuous Activity | 7 | 14 | 21
Primary Tumor [Number; unit: participants]
  Extrahepatic Bile Duct | 8 | 11 | 19
  Intrahepatic Bile Duct | 14 | 14 | 28
  Gallbladder | 15 | 17 | 32
  Papilla | 4 | 0 | 4
Tumor Histological Type [Number; unit: participants]
  Adenocarcinoma | 39 | 41 | 80
  Adenosquamous Cancer | 2 | 1 | 3
Body Surface Area [Mean (Standard Deviation); unit: square meter (m^2)] | 1.555 (0.195) | 1.523 (0.158) | 1.539 (0.177)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 159.80 (8.75) | 156.67 (8.62) | 158.21 (8.77)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 54.97 (12.31) | 53.91 (9.50) | 54.43 (10.92)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Alive at 1 Year (1-Year Survival Rate)
Description: Percentage of patients alive at 1 year.
Time Frame: 1 year
Population: Number of patients who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Gemcitabine + Cisplatin | Gemcitabine
Number analyzed (Participants) | 41 | 42
percentage of participants | 39 | 31

2. Secondary Outcome: Tumor Response
Description: Response Evaluation Criteria In Solid Tumors - define when cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progression") during treatments. Complete response (CR) = disappearance of all target lesions; Partial Response (PR) = 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) = 20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD) = small changes that do not meet above criteria.
Time Frame: baseline to measured progressive disease (up to 2 years)
Population: Number of patients who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Gemcitabine + Cisplatin | Gemcitabine
Number analyzed (Participants) | 41 | 42
participants
  Complete Response | 0 | 0
  Partial Response | 8 | 5
  Stable Disease | 20 | 16
  Progressive Disease | 9 | 17
  Not Evaluable | 4 | 4
Statistical Analysis 1: Comparison: Gemcitabine + Cisplatin vs Gemcitabine; Test type: Superiority or Other; p = 0.380, Fisher Exact — P-value for response (Complete Response + Partial Response)

3. Secondary Outcome: Progression Free Survival
Description: The period from study entry until disease progression, death or date of last contact.
Time Frame: baseline to measured progressive disease (up to 2 years)
Population: Number of patients who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine + Cisplatin | Gemcitabine
Number analyzed (Participants) | 41 | 42
months | 5.8 [4.1 to 8.2] | 3.7 [2.1 to 5.3]
Statistical Analysis 1: Comparison: Gemcitabine + Cisplatin vs Gemcitabine; Test type: Superiority or Other; p = 0.074, Log Rank

4. Other Pre Specified Outcome: Survival Time
Description: Data of patients lost to follow-up were censored at the last date of confirmation of their survival.
Time Frame: baseline to date of death due to any cause (up to 2 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine + Cisplatin | Gemcitabine
Number analyzed (Participants) | 41 | 42
months | 11.2 [9.1 to 12.5] | 7.7 [6.1 to 11.0]
Statistical Analysis 1: Comparison: Gemcitabine + Cisplatin vs Gemcitabine; Test type: Superiority or Other; p = 0.136, Log Rank

ADVERSE EVENTS:
Arm/Group | Gemcitabine + Cisplatin | Gemcitabine
Serious Adverse Events (participants affected / at risk) | 9/41 | 17/42
Other Adverse Events (participants affected / at risk) | 41/41 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + Cisplatin (N=41) | Gemcitabine (N=42)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 4 (4) | 8 (19)
Haemobilia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 2 (2) | 4 (4)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 2 (3) | 0 (0)
Stent occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (10)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (7)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + Cisplatin (N=41) | Gemcitabine (N=42)
Anaemia (Blood and lymphatic system disorders) | 4 (6) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (3) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 4 (6)
Ascites (Gastrointestinal disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 15 (30) | 14 (17)
Diarrhoea (Gastrointestinal disorders) | 13 (31) | 11 (20)
Nausea (Gastrointestinal disorders) | 28 (100) | 18 (54)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 5 (6)
Vomiting (Gastrointestinal disorders) | 20 (50) | 10 (26)
Fatigue (General disorders) | 24 (67) | 21 (104)
Malaise (General disorders) | 7 (11) | 6 (10)
Oedema (General disorders) | 1 (2) | 6 (7)
Oedema peripheral (General disorders) | 4 (5) | 5 (5)
Pyrexia (General disorders) | 18 (28) | 25 (88)
Cholangitis (Hepatobiliary disorders) | 3 (3) | 5 (5)
Nasopharyngitis (Infections and infestations) | 7 (10) | 11 (15)
Alanine aminotransferase increased (Investigations) | 21 (34) | 22 (67)
Aspartate aminotransferase increased (Investigations) | 22 (35) | 22 (74)
Blood albumin decreased (Investigations) | 9 (16) | 22 (49)
Blood alkaline phosphatase increased (Investigations) | 13 (18) | 17 (29)
Blood amylase increased (Investigations) | 3 (3) | 3 (4)
Blood bilirubin increased (Investigations) | 8 (13) | 12 (18)
Blood chloride decreased (Investigations) | 6 (13) | 5 (6)
Blood cholesterol decreased (Investigations) | 0 (0) | 3 (3)
Blood cholinesterase decreased (Investigations) | 3 (3) | 2 (2)
Blood creatinine increased (Investigations) | 8 (30) | 6 (8)
Blood glucose increased (Investigations) | 5 (8) | 5 (6)
Blood lactate dehydrogenase increased (Investigations) | 15 (30) | 15 (37)
Blood potassium decreased (Investigations) | 7 (17) | 4 (5)
Blood potassium increased (Investigations) | 7 (27) | 6 (24)
Blood sodium decreased (Investigations) | 13 (35) | 8 (11)
Blood urea increased (Investigations) | 5 (20) | 9 (19)
C-reactive protein increased (Investigations) | 11 (17) | 22 (40)
Creatinine renal clearance decreased (Investigations) | 5 (19) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 19 (32) | 21 (47)
Glucose urine present (Investigations) | 3 (6) | 4 (12)
Haematocrit decreased (Investigations) | 24 (41) | 23 (48)
Haemoglobin decreased (Investigations) | 35 (69) | 36 (94)
Neutrophil count decreased (Investigations) | 34 (164) | 29 (115)
Neutrophil count increased (Investigations) | 10 (15) | 16 (27)
Platelet count decreased (Investigations) | 33 (167) | 32 (125)
Platelet count increased (Investigations) | 5 (14) | 19 (54)
Protein total decreased (Investigations) | 9 (26) | 16 (28)
Protein urine present (Investigations) | 11 (20) | 11 (20)
Red blood cell count decreased (Investigations) | 31 (52) | 33 (55)
Weight decreased (Investigations) | 13 (18) | 13 (16)
Weight increased (Investigations) | 5 (10) | 5 (5)
White blood cell count decreased (Investigations) | 36 (153) | 29 (122)
White blood cell count increased (Investigations) | 12 (22) | 23 (39)
White blood cells urine positive (Investigations) | 1 (1) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 33 (110) | 26 (66)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (6) | 5 (5)
Dizziness (Nervous system disorders) | 1 (1) | 5 (7)
Dysgeusia (Nervous system disorders) | 4 (5) | 3 (3)
Headache (Nervous system disorders) | 4 (5) | 7 (16)
Hypoaesthesia (Nervous system disorders) | 4 (4) | 2 (2)
Haematuria (Renal and urinary disorders) | 7 (21) | 8 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (11) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (4)
Rash (Skin and subcutaneous tissue disorders) | 11 (15) | 9 (10)
Bile duct stent insertion (Surgical and medical procedures) | 5 (5) | 8 (10)
Catheter placement (Surgical and medical procedures) | 5 (14) | 12 (35)
Angiopathy (Vascular disorders) | 3 (11) | 3 (4)
Hypertension (Vascular disorders) | 0 (0) | 3 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days